CLINICAL TRIAL: NCT07349264
Title: Boswellia Serrata, Curcumin, and Methylsulfonylmethane Combination Supplementation Improves Joint Health
Brief Title: Flexy3 Supplementation and Joint Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NXTVSION SDN. BHD. (Industry)
Collaborators: UCSI University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Flexy3-Protocol-0001
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Joint; Joint Diseases
Keywords: Arthritis; Boswellia serrata; Curcumin; Methylsulfonylmethane; Quality of Life
MeSH Terms: conditions — Joint Diseases; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Flexy3) (Experimental): The intervention supplement is made in vega capsule form (OriactivTM, Flexy3, Malaysia). Each capsule (500mg) consisted of B. serrata gum extract (100mg), Curcuma Longa (Turmeric) rhizome extract (150mg) and MSM (250mg). Participants were instructed to take two capsules twice daily.
  Interventions: Dietary Supplement: Flexy3 Supplement (OriactivTM, Flexy3, Malaysia)
- Placebo Arm (Placebo Comparator): The placebo consisted of capsules containing only excipients and food coloring, formulated to match the appearance of the active supplement. Participants were instructed to take two capsules twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Flexy3 Supplement (OriactivTM, Flexy3, Malaysia) — Each capsule (500mg) consisted of B. serrata gum extract (100mg), Curcuma Longa (Turmeric) rhizome extract (150mg) and MSM (250mg).
  Arms: Interventional Arm (Flexy3)
Other: Placebo — The placebo consisted of capsules containing only excipients and food coloring, formulated to match the appearance of the active supplement.
  Arms: Placebo Arm

SUMMARY:
The prevalence of osteoarthritis (OA) of the knee, hip, and hand has been estimated at 20% to 30% in the adult population (Neogi and Zhang, 2012). Knee OA is the most common form with prevalence increases throughout the lifespan (Wallace et al., 2017, Nguyen et al., 2011). Globally, knee and hip OA were estimated to be the 11th greatest contributors to years of life lived with disability in 2010 (Cross et al., 2014). On the other hand, rheumatoid arthritis (RA) has been reported to affect 0.1-2.0% of the population worldwide (Almutairi et al., 2021). As with any disease, identifying novel treatment options for managing arthritis and promoting joint health requires an understanding of the underlying etiology that leads to the development of the observed symptoms (Guo et al., 2018, Sandell, 2012). The pathophysiology of cartilage degradation in arthritis is multifactorial, primarily driven by pro-inflammatory cytokines and oxidative stress, and further exacerbated by metabolic comorbidities. (e.g., obesity, diabetes) (Rahmati et al., 2017, Markovics et al., 2021).

In vitro evidence suggests that some natural products may possess anti-inflammatory and anti-oxidative properties and may inhibit the release of key osteoarthritis-related cytokines. There is, therefore, ongoing interest in identifying natural products that safely promote joint health and treat osteoarthritis. Numerous plant extracts, including curcumin, Boswellia extract, and pycnogenol, have shown effect sizes (ES) for reducing pain and functional disability larger than those observed with analgesics and products such as glucosamine and chondroitin (Henrotin and Mobasheri, 2018). A recent literature review and meta-analysis conducted by Liu et al. (2018) reported that a number of natural products produced clinically important effect sizes (ES) of -1.2 to - 1.6 in randomized, controlled trials (RCTs), that exceed what has been observed with traditional OA treatments such as glucosamine and chondroitin, which showed no or small effects (ES = - 0.28 to - 0.34) (Liu et al., 2018a, Liu et al., 2018b).

Boswellia serrata is a tree that is widely distributed in India, and its oily gum resin has traditionally been used for centuries in humans as a remedy to treat inflammatory diseases (Siddiqui, 2011). The resinous part of Boswellia serrata possesses monoterpenes, diterpenes, triterpenes, tetracyclic triterpenic acids and four major pentacyclic triterpenic acids, i.e., β-boswellic acid, acetyl-β-boswellic acid (AβBA), 11-keto-β-boswellic acid and acetyl-11-keto-β-boswellic acid (AKBA) (Al-Yasiry and Kiczorowska, 2016). Boswellic acids with the characteristic pentacyclic triterpene ring can exhibit actions related to the inflammatory cascade, with AKBA being more active, selectively inhibiting a branch of the arachidonic acid cascade (5 LOX) related to the production of leukotrienes without affecting other activities of LOX and COX. The inhibition of 5 LOX and leukotriene synthesis reduces the levels of pro-inflammatory cytokines, leading to decreased cartilage destruction and inflammatory cell chemotaxis and producing a balance in favour of cartilage regeneration (Ammon, 2006, Ammon, 2010).

Boswellia serrata has garnered significant attention for its potential anti-inflammatory and joint-supporting properties. Despite its growing popularity as a supplement, there is a need for more robust, evidence-based research to establish its efficacy in improving joint health. By studying the effects of Boswellia serrata supplementation, this research aims to address gaps in the existing literature, and contribute to the development of effective, natural interventions for individuals experiencing joint discomfort and impaired mobility.

ELIGIBILITY:
Inclusion Criteria:

* Subject with the complains of either pain or stiffness on joint, difficulty in walking and dressing due to arthritis or joint problem that interfered work/daily routine or social activities in the past 3 months
* At least 2/10 on pain scores using visual analogue scale (VAS)
* Age 18 or above
* Willing to comply with interventional plan and comes to do follow up
* Willing to gives consent

Exclusion Criteria:

* Use of any NSAIDS in the last 48 hours
* Use of any Intramuscular/intra-articular/systemic corticosteroid in the last 30 days
* Use of any supplements targeting joint health in the last 30 days
* Significant trauma to knees, including arthroscopy or significant injury to ligaments or menisci of the knee in the last 3 months
* Subject who is currently on medication
* Subject with chronic diseases, including but not limited to hypertension, diabetes, cancer, cardiovascular diseases, chronic respiratory diseases, neurological conditions.
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Inflammation Levels | Week 0, 4, 8 and 12
  Inflammation levels was determined through the biomarkers Matrix Metalloproteinase 8 (MMP-8) , interleukin-1 beta (IL-1b) and tumour necrosis factor-alpha (TNF-a). The levels of interleukin-1 beta (IL-1b) and tumour necrosis factor-alpha (TNF-a) were assayed using ELISA MAX™ Deluxe Set Human IL-1β and ELISA MAX™ Deluxe Set Human TNF-α (BioLegend, Inc) respectively. The level of matrix metalloproteinase 8 (MMP-8) was measured using human MMP-8(Matrix Metalloproteinase 8) ELISA Kit (Elabscience Biotechnology Co., Ltd., Houston, TX, USA)
Severity and Symptoms of Arthritis | Week 0, 4, 8 and 12
  Severity and symptoms of arthritis was measured using Western Ontario and McMaster Universities Osteoarthritis Index. The WOMAC Index is a validated, self-administered questionnaire designed to assess three dimensions of joint health: pain (five items), stiffness (two items), and physical function (16 items).

SECONDARY OUTCOMES:
Standardized health-related quality of life (HRQoL) | Week 0, 4, 8 and 12
  Quality of life was determined using EQ-5D-5L. The EQ-5D-5L is a standardized instrument for measuring health-related quality of life. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each rated on five levels of severity (no problems, slight problems, moderate problems, severe problems, extreme problems).

CONTACTS AND LOCATIONS:
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request. Additional docu-ments including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following pub-lication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Wolfe F. Determinants of WOMAC function, pain and stiffness scores: evidence for the role of low back pain, symptom counts, fatigue and depression in osteoarthritis, rheumatoid arthritis and fibromyalgia. Rheumatology (Oxford). 1999 Apr;38(4):355-61. doi: 10.1093/rheumatology/38.4.355. PMID 10378714
- [Result] Siwach SB, Yadav DR, Arora B, Dalal S, Jagdish. Acute aluminum phosphide poisoning--an epidemiological, clinical and histo-pathological study. J Assoc Physicians India. 1988 Oct;36(10):594-6. No abstract available. PMID 3220807